CLINICAL TRIAL: NCT04839783
Title: Multi-center, Prospective, Single Position, Spine Surgery Outcomes Registry
Brief Title: Single Position Spine Surgery Registry
Acronym: SPSG Registry
Status: Terminated | Type: Observational
Why Stopped: Previously allocated resources had to be redirected, at multiples sites.
Sponsor: Spine and Scoliosis Research Associates (Other)
Responsible Party: Sponsor
Other Study IDs: 20201713
Record Dates: First submitted 2021-03-10; First posted 2021-04-09 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Spine Fusion; Spinal Stenosis; Degenerative Disc Disease
MeSH Terms: conditions — Spinal Stenosis; Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to systematically, prospectively compare surgical fusion techniques for thoracolumbar spinal fusion patients and assess long-term patient outcomes and revision rates following surgery.

DETAILED DESCRIPTION:
The goal of this study is to understand how the difference in positioning of a patient intraoperatively, as part of performing an anterior posterior spine fusion surgery, can affect short term and long term outcomes. This will be accomplished through observational techniques that will not affect the care patients will receive for their spinal conditions.

Patients will be asked to complete health and wellness surveys before and after survey to determine how they are doing before surgery and then what if any changes their respective surgeries have had on their lives. Further spine x-rays that they have taken to plan their surgeries and assess their recovery will be measured, when available. X-rays will not be taken only for research purposes. Additionally aspects of their surgeries will be noted such as where hardware is placed and how long different parts of the surgery took.

Follow-up is planned to be out to 10 years post-operatively with the goal of collecting information about any revision spine surgeries that would happen during those 10 years as well.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years
2. Ability to speak and read comfortably in English
3. Affliction by a spinal condition warranting evaluation for operative treatment

Exclusion Criteria:

1. Current incarceration
2. Individuals incapable of consenting and/or objectively responding to surveys, irrespective of reasonable assistance
3. Women currently pregnant or expecting to become pregnant in the near future
4. Subjects participating in another research study, whose protocol would conflict with comprehensive participation in this study
5. Subjects with psychiatric pathology which may impair judgement or the ability to give informed consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from spinal conditions for which a spine surgeon has recommended an anterior posterior fusion, who meet all inclusion and no exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2025-07-07 (Actual); Study Completion 2025-07-07 (Actual)

PRIMARY OUTCOMES:
Difference in Patient-Reported Outcomes Measurement Information System (PROMIS) Domain-Pain Interference | 10 years
  Assess the difference between pre-op and post-op scores. Scores range from 0-100. A higher number indicates more Pain Interference.
Difference in Patient-Reported Outcomes Measurement Information System (PROMIS) Domain-Pain Intensity | 10 years
  Assess the difference between pre-op and post-op scores. Scores range from 0-100. A higher number indicates more Pain Intensity.
Difference in Patient-Reported Outcomes Measurement Information System (PROMIS) Domain-Depression | 10 years
  Assess the difference between pre-op and post-op scores. Scores range from 0-100. A higher number indicates more Depression.
Difference in Patient-Reported Outcomes Measurement Information System (PROMIS) Domain-Anxiety | 10 years
  Assess the difference between pre-op and post-op scores. Scores range from 0-100. A higher number indicates more Anxiety.
Difference in Patient-Reported Outcomes Measurement Information System (PROMIS) Domain-Physical Function Scores | 10 years
  Assess the difference between pre-op and post-op scores. Scores range from 0-100. A higher number indicates less Physical Function.
Difference in Radiographic Measurements-Cobb Angles | 10 years
  Assess the difference between pre-op and post-op measurements of Cobb Angles using available spinal x-rays for patients whose Cobb Angle was to be changed as part of their surgical plan.
Difference in Radiographic Measurements-Fractional Curve Cobb Angles | 10 years
  Assess the difference between pre-op and post-op measurements of Fractional Curve Cobb Angles using available spinal x-rays for patients whose Fractional Curve Cobb Angle was to be changed as part of their surgical plan.
Difference in Radiographic Measurements-C7 Sagittal Vertical Alignment (SVA) | 10 years
  Assess the difference between pre-op and post-op measurements of C7 SVA using available spinal x-rays for patients whose C7 SVA was to be changed as part of their surgical plan.
Difference in Radiographic Measurements-Coronal Sagittal Vertical Alignment (SVA) | 10 years
  Assess the difference between pre-op and post-op measurements of Coronal SVA using available spinal x-rays for patients whose Coronal SVA was to be changed as part of their surgical plan.
Difference in Radiographic Measurements-Pelvic Incidence (PI) | 10 years
  Assess the difference between pre-op and post-op measurements of PI using available spinal x-rays for patients whose PI was to be changed as part of their surgical plan.
Difference in Radiographic Measurements-Pelvic Tilt (PT) | 10 years
  Assess the difference between pre-op and post-op measurements of spinal x-rays for patients whose PT was to be changed as part of their surgical plan.
Difference in Radiographic Measurements-Lumbar Lordosis (LL) | 10 years
  Assess the difference between pre-op and post-op measurements of spinal x-rays for patients whose LL was to be changed as part of their surgical plan.
Difference in Radiographic Measurements-T1 Pelvic Angle (TPA) | 10 years
  Assess the difference between pre-op and post-op measurements of spinal x-rays, for patients whose TPA was to be changed as part of their surgical plan.
Revision Incidence | 10 years
  Determine the incidence of spine surgery revisions after the initial surgery.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (5):
  - New England Baptist Hospital, Boston, Massachusetts
  - NYU Langone Health, New York, New York
  - Atlantic Neurosurgical and Spine Specialists, Wilmington, North Carolina
  - The Spine Clinic of Oklahoma City, Oklahoma City, Oklahoma
  - Austin Spine, Austin, Texas
- Melbourne Orthopedic Group, Windsor, Victoria, Australia